CLINICAL TRIAL: NCT03826225
Title: Cardiac Monitor Employee Study
Acronym: CARMEL
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CARMEL
Record Dates: First submitted 2019-01-24; First posted 2019-02-01 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Cohort: All participants are considered to be in the study cohort and will have the study device placed externally on their skin in order to collect human ECG data.

SUMMARY:
This purpose of this study is to collect ECG data from a wearable cardiac monitor in order to evaluate end-to-end performance of a cardiac monitor system and associated data management accessories.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the usability of the Wearable Cardiac Monitor (WCM) system including the WCM, Mobile Monitors (patient and clinician), Magnet and LATITUDE Clarity(TM) Server. The study will exercise the end-to-end system utilizing human ECG data generated by the wearable cardiac monitor.

ELIGIBILITY:
Inclusion Criteria:

* Willing and capable to provide informed consent
* Age 18 or above
* Employee of the study sponsor
* Willing and able to follow protocol requirements

Exclusion Criteria:

* Currently enrolled in another clinical study that interferes with data collection
* Currently implanted with an active medical electronic device
* Known allergies to the materials that may come in contact with the skin
* Any active skin condition on the chest reported by the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll volunteer adult participants who are employees of the study sponsor and who meet all eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Evaluate WCM System End-To-End Performance | 3 months
  Characterize rate of success of wireless data transmissions from wearable cardiac monitor to LATITUDE Clarity(TM) server

CONTACTS AND LOCATIONS:
Overall Officials: Dave Perschbacher, Principal Investigator — Senior R&D Fellow
Locations (1):
- Boston Scientific, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No